CLINICAL TRIAL: NCT00144651
Title: An Open-label, Extension, Phase II Study to Evaluate the Long-term Safety and Efficacy of MRA in Patients With RA Who Were Participated in Study MRA009JP
Brief Title: Study of MRA in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA010JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MRA(Tocilizumab)

INTERVENTIONS:
Drug: MRA(Tocilizumab) — 8mg/kg/4 weeks for 1 year

SUMMARY:
This is an open-label, extension, Phase II study to evaluate the long-term safety and efficacy of MRA in Patients with RA who were participated in Study MRA009JP.

ELIGIBILITY:
Inclusion Criteria:

* Patients administered MRA more than 2 times in preceding study, MRA009JP, and evaluated the efficacy and the safety.
* Patients confirmed to have shown the safety in the preceding study.

Exclusion Criteria:

* Patients with Class IV Steinbrocker functional activity at evaluation within 4 weeks before treatment with the study drug
* Patients who received any of the following treatments between the start of preceding study and the registration of this study.

  1. Plasma exchange therapy
  2. Surgical treatment (e.g., operation)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2001-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
ACR 20% responder rate compared to the pre-treatment in the preceding study | throughout study
Frequency and severity of adverse events and adverse drug reactions | week0,week4,week8,week12,and LOBS

SECONDARY OUTCOMES:
Time course of DAS28,compared to the pre-treatment in the preceding study | week 0,week 4,week 8,week 12, LOBS
Time course of the ACR 20%, 50%, and 70% responder rates compared to the pre-treatment in the preceding study | week 0,week 4,week 8,week 12, LOBS
ACR N AUC compared to the pre-treatment in the preceding study | week 0,week 4,week 8,week 12, LOBS
Time course of the ACR core set variables compared to the pre-treatment in the preceding study | week 0,week 4,week 8,week 12, LOBS

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical